CLINICAL TRIAL: NCT06119867
Title: Comparison Between the European and Japanese Pathological Investigation for Colon Cancer (SPACE)
Acronym: SPACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Principal Investigator, Vladimir Balaban, Principal Investigator, Russian Society of Colorectal Surgeons
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0004
Record Dates: First submitted 2023-10-12; First posted 2023-11-07 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Japanese pathological investigation method group (Experimental): The surgeon will be involved into the Japanese pathological investigation method. The surgeon will perform the intraoperative markings and the postoperative lymph node harvest, after which the specimen will be assessed by the pathologist.
  Interventions: Procedure: Japanese pathological investigation
- European pathological investigation method group (Active Comparator): After receiving the resected specimen, the entire process will be independently managed by the pathologist.
  Interventions: Procedure: European pathological investigation

INTERVENTIONS:
Procedure: Japanese pathological investigation — Japanese pathological investigation
  Arms: Japanese pathological investigation method group
Procedure: European pathological investigation — The European pathology evaluation method involves the analysis of fresh and intact specimens. Pathologists carefully inspect the entire specimen's appearance and assess the surgical resection plane and capture complete photographs for documentation purposes before further sectioning the specimen. During specimen processing, the CRM is initially marked with ink or other markers. After fixation, macroscopic data are recorded, and the entire length of the intestine is cut into cross-sections at intervals of 3-4 millimeters. These sections are then undergoing subsequent systematic pathological examination. However, the surgeon will be involved in the Japanese pathological investigation method. Intraoperative markings will be made 10 cm bilaterally from the primary tumor area. The resected colon will be incised at 1 cm intervals, after which the pericolic lymph nodes will be harvested. Each single retrieved lymph node will be packed up independently and will be examined by the pathologist.
  Arms: European pathological investigation method group

SUMMARY:
In general, the European pathological examination method primarily relies on pathologists and does not require the involvement of surgeons. The Japanese pathological evaluation approach, on the other hand, involves the intervention of surgeons, particularly in the extraction of lymph nodes from fresh specimens and the assessment of specimen quality. Given that the Japanese pathological assessment method lacks systematic evaluation and there is currently no literature clearly demonstrating its diagnostic accuracy, the main objective of this study is to verify whether the diagnostic accuracy of the Japanese pathological investigation method is inferior to that of the European pathological evaluation method.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colon cancer who underwent colectomy;
* Patients with pathological confirmed adenocarcinoma;
* Patients agreed to participate in the study.

Exclusion Criteria:

* Patients suffered from rectal cancer;
* Patients diagnosed with colon cancer but did not undergo colectomy;
* Patients refused participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparision of the incidence of stage III colon cancer between European and Japanese pathological investigation methods. | up to 24 months
  indentification of the rate of postive lymph nodes

SECONDARY OUTCOMES:
The role of immunohistochemical examination in the Node (N) stage determination | up to 24 months
  indentification of the rate of postive lymph nodes using immunohistochemical examination
Comparison of the lymph node ratio (LNR) between the European and Japanese pathological approaches | up to 24 months
  LNR=Postivie lymph node/ Total retrived lymph node
Comparison of the pT Stage between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of the pathological T stages
Comparison of the resection margin (proximal, distal, circular) between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of the postive proximal, distal or circular resection margin
Comparison of the tumor budding between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of tumor budding
Comparison of the tumor-infiltrating lymphocytes (TIL) count between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of the tumor-infiltrating lymphocytes (TIL) count
Comparison of the extracapsular invasion between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of the extracapsular invasion
Comparison of the extramural invasion (venous, lymphatic, perineural) between the European and Japanese pathological approaches | up to 24 months
  indentification of the rate of the venous, lymphatic or perineural extramural invasion

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Balaban, Principal Investigator — Sechenov University; Petr Tsarkov, Study Director — Sechenov University
Locations (1):
- Clinic of coloproctology and minimally invasive surgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No